CLINICAL TRIAL: NCT05821504
Title: Effects of Plyometric- and Cycle-Based High-Intensity Interval Training on Body Composition, Aerobic Capacity, and Muscle Function in Young Females: a Field-based Group Fitness Assessment
Brief Title: High-Intensity Interval Training and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Principal Investigator, Garrett Hester, Associate Professor of Exercise Science, Kennesaw State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0465
Record Dates: First submitted 2023-03-14; First posted 2023-04-20 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two groups performed different types of high-intensity interval training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric High-Intensity Interval Training (Experimental): This group performed high-intensity interval training consisting of body-weight, plyometric exercises involving jumping.
  Interventions: Behavioral: High-Intensity Interval Training
- Cycling High-Intensity Interval Training (Experimental): This group performed high-intensity interval training consisting of cycling exercise.
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — The training intervention is a popular exercise format that consist of alternating brief bouts of high-intensity efforts with bouts of light effort or complete rest.

SUMMARY:
The goal of this clinical trial was to compare to different types of high-intensity interval training in young, healthy females. The main questions were: Will changes in body composition differ between the two interventions? Will changes in endurance and muscle performance differ between the two interventions? Participants were randomized to 8 weeks of high-intensity interval training involving body weight, plyometric exercises or cycling only. Researchers compared changes in endurance performance, body composition, and muscle performance to determine if there were differences between groups.

DETAILED DESCRIPTION:
The purpose of this study was to compare the effects of plyometric- and cycle-oriented high-intensity interval training on body composition, aerobic capacity, and skeletal muscle size, quality, and function in recreationally trained females. Young (21.7 ± 3.1 yrs), recreationally active females were randomly assigned to 8 weeks of twice weekly plyometric (n = 15) or cycling (n = 15) high-intensity interval training. The plyometric-oriented Les Mills BODYATTACK program was used for the plyometric group whereas Les Mills SPRINT, which exclusively involves stationary cycling, represented the cycling group. Both protocols involved alternating high-intensity and recovery intervals, and participants were consistently instructed to give maximal effort during the 'work' periods.

The 30 min plyometric routines included four blocks of high-intensity exercise intervals. The 'work' portions consisted of the following exercises: high-knee runs, plyometric lunges, jumping jacks, squat jumps, burpees, and speed-agility patterns. The recovery periods consisted of complete rest (transitioning between exercises), a light jog, or a low impact stepping motion. On average, participants were instructed to give maximal effort for 1-2 min, with recovery intervals of 15-45 sec. Four separate routines were used throughout the duration of the study, keeping one routine per week; participants completed each routine a total of 4 times within a session.

The 30 min cycling routines were performed on upright stationary bikes (Schwinn, AC Performance, Chicago, IL). Protocols involved 'work' ranging from 20-80 sec with recovery intervals between 10-60 sec. Recovery intervals consisted of complete rest on bike or particularly slow cycling. Resistance and cycling speed were relatively variable across sessions, with some intervals of higher resistance and lower speed and others involving lower resistance and higher speed (e.g., >120 RPMs). The same four workouts were used throughout the duration of the study alternating each week.

Body composition (4-compartment model), VO2peak, countermovement jump performance, muscle size and echo intensity (muscle quality) as well as strength and power of the knee extensors and plantar flexors were measured before and after training. Body composition testing was completing using dual-energy x-ray absorpiometry, air displacement plethysmogrphay, and bioeletrical impedance. VO2peak was measured using a standardized maximal exercise test on a treadmill. Countermovement jump height and power was recorded with participants performing jumps on a force plate. Muscle size and quality were determined using non-invasive ultrasonography. Finally, serum growth hormone responses to the VO2peak test were measured before and after the protocols.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-35 years of age
* Female
* Currently participating in 2-4 days of structured exercise for 30-75 minutes for the last 6 months

Exclusion Criteria:

* Currently participating in these exercise formats (2x/week within last 3 months)
* Engaging in high intensity interval training for more than 30 min/week
* Have diagnosed disorders/diseases in the following: cardiovascular, pulmonary, immunological, or metabolic
* Current musculoskeletal injuries
* Pregnant or think you may be pregnant
* Currently taking any non-steroidal anti-inflammatory drug(s) or steroidal drug(s)
* Currently a smoker or has consistently smoked within the last year
* Has a positive written or verbal pre-study drug screen including alcohol (more than 7 drinks/week), THC/cannabinoids, amphetamines, benzodiazepines, cocaine, opioids, phencyclidine, barbiturates, cotinine.
* Currently taking any medication that will significantly affect your heart rate response to exercise
* If you miss four or more classes, you will be excluded from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Muscle composition at baseline | Pre-intervention
  echo-intensity value derived from ultrasound that indicates the amount of fat infiltration in muscle
Muscle composition after 8-week intervention | At week 9
  echo-intensity value derived from ultrasound that indicates the amount of fat infiltration in muscle

SECONDARY OUTCOMES:
Fat mass at baseline | Pre-intervention
  Amount of fat tissue a person possesses
Fat mass after 8-week intervention | At week 9
  Amount of fat tissue a person possesses
Group average growth hormone response (concentration at microLiters/Liters) at baseline | Pre-intervention
  The acute, exercise-induced response for growth hormone
Group average growth hormone response (concentration at microLiters/Liters) after 8-week intervention | At week 9
  The acute, exercise-induced response for growth hormone
Countermovement jump height at baseline | Pre-intervention
  Height of jump
Countermovement jump height after 8-week intervention | At week 9
  Height of jump
Time to peak torque at baseline | Pre-intervention
  How quickly muscle torque is generated
Time to peak torque after 8-week intervention | At week 9
  How quickly muscle torque is generated
Maximal oxygen consumption at baseline | Pre-intervention
  Standard measure of maximal oxygen consumption or peak aerobic capacity during exercise
Maximal oxygen consumption after 8-week intervention | At week 9
  Standard measure of maximal oxygen consumption or peak aerobic capacity during exercise
Body fat percentage at baseline | Pre-intervention
  Relative amount of body fat a person possesses
Body fat percentage after 8-week intervention | At week 9
  Relative amount of body fat a person possesses
Fat-free mass at baseline | Pre-intervention
  Amount of non-fat tissue a person possesses
Fat-free mass after 8-week intervention | At week 9
  Amount of non-fat tissue a person possesses
Peak torque at baseline | Pre-intervention
  Strength of a muscle
Peak torque after 8-week intervention | At week 9
  Strength of a muscle
Muscle cross-sectional area at baseline | Pre-intervention
  The size of a muscle
Muscle cross-sectional area after 8-week intervention | At week 9
  The size of a muscle
Muscle power at baseline | Pre-intervention
  Product of torque and velocity as determined on a dynamometer
Muscle power after 8-week intervention | At week 9
  Product of torque and velocity as determined on a dynamometer

OTHER OUTCOMES:
Weekly exercising heart rate | during 8-week exercise intervention
  A descriptor of the exercise physiological intensity for both protocols
Weekly exercising perceived effort | during 8-week exercise intervention
  Perceived intensity derived from the rating of perceived exertion scale
Calorie consumption at baseline | Pre-intervention
  Amount of calories consumed at beginning and end of protocol
Calorie consumption after 8-week intervention | At week 9
  Amount of calories consumed at beginning and end of protocol
Protein consumption at baseline | Pre-intervention
  Amount of protein consumed at beginning and end of protocol
Protein consumption after 8-week intervention | At week 9
  Amount of protein consumed at beginning and end of protocol
Peak heart during maximal testing at baseline | Pre-intervention
  The highest heart rate attained during maximal exercise testing
Peak heart during maximal testing after 8-week intervention | At week 9
  The highest heart rate attained during maximal exercise testing

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share.

REFERENCES:
- [Derived] Holmes AJ, Stratton MT, Bailly AR, Gottschall JS, Feito Y, Ha PL, Lavigne A, Persaud K, Gagnon HL, Krueger A, Modjeski A, Esmat TA, Harper LN, VanDusseldorp TA, Hester GM. Effects of plyometric- and cycle-based high-intensity interval training on body composition, aerobic capacity, and muscle function in young females: a field-based group fitness assessment. Appl Physiol Nutr Metab. 2023 Dec 1;48(12):932-945. doi: 10.1139/apnm-2022-0465. Epub 2023 Aug 9. PMID 37556856